CLINICAL TRIAL: NCT06175988
Title: Adiposité Viscérale, Tonus Vagal Et Préférences Alimentaires : Une Étude Pilote
Brief Title: Visceral Adiposity, Vagal Tone and Food Preferences: a Pilot Study
Acronym: ObVague
Status: Recruiting | Type: Observational
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Sylvain Iceta, Principal Investigator, Laval University
Other Study IDs: 2024-4097, 22392
Record Dates: First submitted 2023-12-01; First posted 2023-12-19 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Adiposity; Food Preferences; Eating Behavior
MeSH Terms: conditions — Obesity; Food Preferences; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Visceral Adiposity: No intervention to be adminstrated. Participants will be considered based on their visceral adiposity (ctageorial and continous). Visceral adiposity index is computed with BMI, waist circumference, triglyceridemia, HDL-cholesterol levels, and biological sex.
  Interventions: Other: Visceral adiposity

INTERVENTIONS:
Other: Visceral adiposity — Visceral adiposity assess by the visceral adiposity index

SUMMARY:
Food preferences are defined by a number of measurable parameters, such as per se food choices, sensitivity of taste and olfactory sensory perceptions, hedonic appreciation of foods ("liking") and motivation to consume them ("wanting"). These food preferences are fundamental to the quality of food intake, and are therefore a key factor influencing weight loss or maintenance of a stable weight. Obesity is also associated with reduced sensory sensitivity to taste and smell, as well as disturbances in the responses of the food reward system.

However, the internal, or physiological, mechanisms impacting these food preferences are still poorly understood. To date, several studies seem to point to the role of body composition, in particular visceral adiposity, or adiposity surrounding the digestive organs. Indeed, a high level of visceral adiposity is associated with the onset of numerous cardiometabolic disorders, but also with altered sensory perceptions.

This relationship could be mediated by the vagus nerve, which connects the digestive organs to the brain, enabling the perception of internal signals sent by the body, such as feelings of hunger or satiety. Low vagal activity is associated not only with abdominal obesity, but also with reduced sensory sensitivity to taste and smell, and changes in food choices in favor of energy-dense foods (rich in fats and/or sugars). Electrical stimulation of the vagus nerve is now recognized as a possible treatment for morbid obesity in the USA, but the mechanisms leading to the expected weight loss are still debated. Similarly, an increase in vagal tone has been found in patients who have undergone bariatric surgery for the treatment of severe complicated to morbid obesity, in parallel with sensory disturbances.

The overall aim of this project is to explore and confirm the relationship between visceral adiposity and various food preference parameters, such as olfactory and gustatory perceptions and reward system responses, involving liking and wanting certain foods and associated behaviors. This project also aims to shed light on the possible mediation of the vagus nerve in this relationship.

ELIGIBILITY:
Inclusion Criteria:

* Have a BMI between 18.5 and 35 kg/m²;
* French-speaking;
* Be able to travel to the Research Center of the Institut Universitaire de Cardiologie et Pneumologie de Québec for an investigative visit.

Exclusion Criteria:

* Smokers ;
* Women who know they are pregnant, breastfeeding or menopausal;
* Who have been diagnosed with type I or type II diabetes;
* Having undergone bariatric surgery or obesity medication (GLP1 analogue, naltrexon-bupropion combination, etc.);
* Presenting an allergy or intolerance to one of the products used in the sensory tests (taste test: sucrose, sodium chloride, citric acid, quinine hydrochloride dihydrate; olfactory test: citrus, lemongrass, cinnamon, mint, peppermint, banana, anise, turpentine, garlic, coffee, apple, clove, pineapple, rose, geranium, eucalyptus, wormwood, fennel, caraway, leather, n-butanol, linalool, pyridine, diethyl phthalate, propylene glycol);
* Have a history of pathologies which, in the investigator's opinion, could interfere with the study criteria, such as ENT, neurological, upper digestive or cardiac pathologies;
* Receiving long-term pharmacological treatment, in particular antidepressants, antipsychotics, benzodiazepines, beta-blockers, etc. ;
* Presenting or having presented in the last 6 months a thymic episode such as depression, bipolar disorder, etc. ;
* Wearing a cardiostimulator (pacemaker);
* Minors or adults under guardianship.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adult men and women aged between 18 and 45 will be selected. This age limitation applied to both sexes will limit the risk of including post-menopausal women, without unbalancing the average age between the biological sexes. We will meet participants during the follicular phase of their cycle (beginning on the first day of menstruation and ending at ovulation).
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
"Taste Strips" total score | Baseline
  Taste identification score for sweet, salty, bitter, and sour (/16). The test used is "Taste Strips" (ODOFIN, Burghart Messtechnik GmbH, Holm, Germany).
TDI score, or "Sniffin Sticks" total score | Baseline
  Olfaction score based on odor detection (Threshold), Discrimination, and Identification (/48). The test used is "Sniffin Sticks" (ODOFIN, Burghart Messtechnik GmbH, Holm, Germany).
"Explicit liking" score for high-fat/sweet foods | Baseline
  "Explicit liking" will be measured using visual analog scales anchored at each end with "not at all" and "extremely" to answer the question "How pleasant would it be to taste this food now?" while seeing pictures of food items. (/100) The task used is the "Leeds Food Preference Questionnaire".
"Explicit liking" score for high-fat/savoury foods | Baseline
  "Explicit liking" will be measured using visual analog scales anchored at each end with "not at all" and "extremely" to answer the question "How pleasant would it be to taste this food now?" while seeing pictures of food items. (/100) The task used is the "Leeds Food Preference Questionnaire".
"Explicit liking" score for low-fat/high-sweet foods | Baseline
  "Explicit liking" will be measured using visual analog scales anchored at each end with "not at all" and "extremely" to answer the question "How pleasant would it be to taste this food now?" while seeing pictures of food items. (/100) The task used is the "Leeds Food Preference Questionnaire".
"Explicit liking" score for low-fat/savoury foods | Baseline
  "Explicit liking" will be measured using visual analog scales anchored at each end with "not at all" and "extremely" to answer the question "How pleasant would it be to taste this food now?" while seeing pictures of food items. (/100) The task used is the "Leeds Food Preference Questionnaire".
"Explicit wanting" score for high-fat/sweet foods | Baseline
  "Explicit wanting" will be measured using visual analog scales anchored at each end with "not at all" and "extremely" to answer the question "How much would like to eat some of this food now?" while seeing pictures of food items. (/100) The task used is the "Leeds Food Preference Questionnaire".
"Explicit wanting" score for high-fat/savoury foods | Baseline
  "Explicit wanting" will be measured using visual analog scales anchored at each end with "not at all" and "extremely" to answer the question "How much would like to eat some of this food now?" while seeing pictures of food items. (/100) The task used is the "Leeds Food Preference Questionnaire".
"Explicit wanting" score for low-fat/sweet foods | Baseline
  "Explicit wanting" will be measured using visual analog scales anchored at each end with "not at all" and "extremely" to answer the question "How much would like to eat some of this food now?" while seeing pictures of food items. (/100) The task used is the "Leeds Food Preference Questionnaire".
"Explicit wanting" score for low-fat/savoury foods | Baseline
  "Explicit wanting" will be measured using visual analog scales anchored at each end with "not at all" and "extremely" to answer the question "How much would like to eat some of this food now?" while seeing pictures of food items. (/100) The task used is the "Leeds Food Preference Questionnaire".
"Implicit wanting" score for high-fat/sweet foods | Baseline
  "Implicit wanting" will be calculated using a forced-choice task. It involves the presentation of successive pairs of food pictures, each pair being the object of a spontaneous preferential choice by the volunteer. A score is calculated from the frequency of choice and non-choice of said category and the reaction time of the participants. This score ranges from -100 to 100 and is interpreted in relation to the scores for the other food categories assessed in the task. A positive score indicates that the food category under consideration was chosen more often and more quickly than the others. A negative score indicates the opposite. The task used is the "Leeds Food Preference Questionnaire".
"Implicit wanting" score for high-fat/savoury foods | Baseline
  "Implicit wanting" will be calculated using a forced-choice task. It involves the presentation of successive pairs of food pictures, each pair being the object of a spontaneous preferential choice by the volunteer. A score is calculated from the frequency of choice and non-choice of said category and the reaction time of the participants. This score ranges from -100 to 100 and is interpreted in relation to the scores for the other food categories assessed in the task. A positive score indicates that the food category under consideration was chosen more often and more quickly than the others. A negative score indicates the opposite. The task used is the "Leeds Food Preference Questionnaire".
"Implicit wanting" score for low-fat/sweet foods | Baseline
  "Implicit wanting" will be calculated using a forced-choice task. It involves the presentation of successive pairs of food pictures, each pair being the object of a spontaneous preferential choice by the volunteer. A score is calculated from the frequency of choice and non-choice of said category and the reaction time of the participants. This score ranges from -100 to 100 and is interpreted in relation to the scores for the other food categories assessed in the task. A positive score indicates that the food category under consideration was chosen more often and more quickly than the others. A negative score indicates the opposite. The task used is the "Leeds Food Preference Questionnaire".
"Implicit wanting" score for low-fat/savoury foods | Baseline
  "Implicit wanting" will be calculated using a forced-choice task. It involves the presentation of successive pairs of food pictures, each pair being the object of a spontaneous preferential choice by the volunteer. A score is calculated from the frequency of choice and non-choice of said category and the reaction time of the participants. This score ranges from -100 to 100 and is interpreted in relation to the scores for the other food categories assessed in the task. A positive score indicates that the food category under consideration was chosen more often and more quickly than the others. A negative score indicates the opposite. The task used is the "Leeds Food Preference Questionnaire".

SECONDARY OUTCOMES:
Standard deviation of the N-N interval (SDNN) | Baseline
  Parameter of the heart rate variability, indirect indicator of the vagal tone (ms). Standard deviation of NN intervals. Measured using a 48 hours Holter monitor.
pNN50 | Baseline
  Parameter of the heart rate variability, indirect indicator of the vagal tone (%). Percentage of successive R-R intervals that differ by more than 50 ms. Measured using a 48 hours Holter monitor.
Root mean square of successive N-N interval difference (RMSSD) | Baseline
  Parameter of the heart rate variability, indirect indicator of the vagal tone (ms). Root mean square of successive R-R interval differences. Measured using a 48 hours Holter monitor.
Low Frequency (LF) | Baseline
  Parameter of the heart rate variability, indirect indicator of the vagal tone (ms²). Power spectral density of low frequencies. Measured using a 48 hours Holter monitor.
High Frequency (HF) | Baseline
  Parameter of the heart rate variability, indirect indicator of the vagal tone (ms²). Power spectral density of high frequencies. Measured using a 48 hours Holter monitor.
LF/HF ratio | Baseline
  Parameter of the heart rate variability, indirect indicator of the vagal tone (a.u.). Measured using a 48 hours Holter monitor.
Sweet Perceived Intensity | Baseline
  Measured during the "Taste Strips" using "9 Likert scales" ranging from "no taste" to "intense" will be used. A score ranging from 1 to 9 will be calculated.
Salty Perceived Intensity | Baseline
  Measured during the "Taste Strips" using "9 Likert scales" ranging from "no taste" to "intense" will be used. A score ranging from 1 to 9 will be calculated.
Bitter Perceived Intensity | Baseline
  Measured during the "Taste Strips" using "9 Likert scales" ranging from "no taste" to "intense" will be used. A score ranging from 1 to 9 will be calculated.
Sour Perceived Intensity | Baseline
  Measured during the "Taste Strips" using "9 Likert scales" ranging from "no taste" to "intense" will be used. A score ranging from 1 to 9 will be calculated.
Sweet Perceived Appreciation | Baseline
  Measured during the "Taste Strips" using "9 Likert scales" ranging from "extremely unpleasant" to "extremely pleasant" will be used. A score ranging from 1 to 9 will be calculated.
Salty Perceived Appreciation | Baseline
  Measured during the "Taste Strips" using "9 Likert scales" ranging from "extremely unpleasant" to "extremely pleasant" will be used. A score ranging from 1 to 9 will be calculated.
Bitter Perceived Appreciation | Baseline
  Measured during the "Taste Strips" using "9 Likert scales" ranging from "extremely unpleasant" to "extremely pleasant" will be used. A score ranging from 1 to 9 will be calculated.
Sour Perceived Appreciation | Baseline
  Measured during the "Taste Strips" using "9 Likert scales" ranging from "extremely unpleasant" to "extremely pleasant" will be used. A score ranging from 1 to 9 will be calculated.
Odors Perceived Intensity | Baseline
  Measured during the "Sniffin Sticks" (identification test) using "9 Likert scales" ranging from "no odor" to "intense" will be used. A score ranging from 1 to 9 will be calculated.
Odors Perceived Appreciation | Baseline
  Measured during the "Sniffin Sticks" (identification test) using "9 Likert scales" ranging from "extremely unpleasant" to "extremely pleasant" will be used. A score ranging from 1 to 9 will be calculated.
Satiety volume as a percentage of total volume (Water Load Task) | Baseline
  Indicator of gastric interoceptive capacities obtained during the "Water Load Task".
Beck Depression Inventory II (BDI-II) score | Baseline
  Evaluates severity of depressive symptoms using a validated questionnaire. Minimum score : 0; Maximun score : 63; Higher scores mean a worse outcome.
State-Trait Anxiety Inventory (STAI) score | Baseline
  Evaluates severity of anxiety symptoms using a validated questionnaire. The questionnaire includes two scales (20 items) consisting of a total of 40 questions. For each scale the minimum score is 0 and the maximun score is 80. Higher scores mean a worse outcome.
Eating Disorder Examination Questionnaire (EDE-Q) score | Baseline
  Evaluates presence of eating disorders using a validated questionnaire. The measure provides four attitudinal subscale scores: Restraint (5 items), Eating Concern (5 items), Shape Concern (8 items), and Weight Concern (5 items). An overall Global score is the mean of the four subscale scores. Responses are on a 7-point ordinal response; minimum score : 0, maximun score: 6; higher scores mean a worse outcome.
Food Craving Trait Questionnaire (FCQ T) score | Baseline
  Evaluates severity of cravings using a validated questionnaire. Minimum : 39; Maximum : 234; Higher scores mean a worse outcome.
Food Craving State Questionnaire (FCQ S) score | Baseline
  Evaluates severity of cravings using a validated questionnaire. Minimum : 15; Maximum : 75; Higher scores mean a worse outcome.
Body Awareness Questionnaire (BAQ) score | Baseline
  Evaluates attention to intern signals (interoception) using a validated questionnaire. Minimum score: 18; Maximun score: 126; Higher scores mean a better outcome.
CCK fasting blood levels | Baseline
  Fasting blood sample. (mmol/L)
PYY fasting blood levels | Baseline
  Fasting blood sample. (mmol/L)
GLP-1 fasting blood levels | Baseline
  Fasting blood sample. (mmol/L)
Glicentine fasting blood levels | Baseline
  Fasting blood sample. (mmol/L)
Oxytomodulin fasting blood levels | Baseline
  Fasting blood sample. (mmol/L)
LPS fasting blood levels | Baseline
  Associated with adipose tissue dysfunction. Fasting blood sample. (mmol/L)
IL-6 fasting blood levels | Baseline
  Associated with adipose tissue dysfunction. Fasting blood sample. (mmol/L)
Fasting Glycemia | Baseline
  Fasting blood sample. (mmol/L)
Fasting Insulinemia | Baseline
  Fasting blood sample. (pmol/L)
Appetite scores | Baseline
  Calculated on the basis of a rating from 0 to 10 for each of the following parameters: sensation of hunger, desire to eat, satiation and prospective consumption. These ratings will be estimated using 100 mm-long visual analog scales annotated with "not at all" and "extremely", on the left and right of the scale respectively, to answer the following questions: "At the moment, how hungry are you?", "At the moment, how hungry are you?", "At the moment, how hungry are you?" and "At the moment, how hungry do you think you are?".
  Before each tests on the exploration day (taste, olfaction, LFPQ, Water Load Task, questionnaires)

CONTACTS AND LOCATIONS:
Locations (1):
- IUCPQ, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided